CLINICAL TRIAL: NCT05468437
Title: Telenutrition to Improve Cardiometabolic Health and Quality of Life Among Individuals With Spinal Cord Injury
Brief Title: Telenutrition for Individuals With SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Clara Valley Health & Hospital System (Other)
Collaborators: San Jose State University (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-038
Record Dates: First submitted 2022-06-21; First posted 2022-07-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Obesity; Cardiometabolic Syndrome
Keywords: Spinal Cord injury; Obesity; Cardiometabolic; cardiovascular; bowel; bladder; nutrition; telehealth
MeSH Terms: conditions — Spinal Cord Injuries; Obesity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: This is a wait-list control study. Individuals in the immediate treatment group will receive the intervention in the first 3 months, followed by a 3 month durability phase. The delayed treatment group will receive the intervention in the second 3 month period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental): Three months of treatment followed by a 3 month durability phase
  Interventions: Behavioral: Telenutrition
- Delayed Treatment (Experimental): A 3 month waitlist period followed by 3 months of treatment
  Interventions: Behavioral: Telenutrition

INTERVENTIONS:
Behavioral: Telenutrition — Nutrition education and individualized nutrition counseling will be done with a Registered Dietitian via video-conferencing with iPad FaceTime, which is aimed to decrease the risk of complications like obesity, high cholesterol, or diabetes, and explore associations between bowel and bladder function and nutrition. The telenutrition counseling consists of 6 sessions that are scheduled approximately 2 weeks apart. The first session will last approximately 1 hour, while sessions 2-6 will last approximately 30mins. During these sessions, the Registered Dietitian will share nutrition education tailored towards people with SCI. You will be involved in developing personal nutrition goals and the dietitian will help you address barriers to meeting your goals and provide individualized feedback to improve and maintain your nutrition. Telenutrition appointments will maintain privacy and will not be recorded.

SUMMARY:
This study will provide nutrition counseling via FaceTime on an iPad to persons with traumatic spinal cord injury (SCI) who are overweight or obese and are at least one-year post-injury. Nutrition counseling may help participants to develop eating behaviors that match the participants' needs and help improve heart health. The purpose of this project is to decrease the risk of complications like obesity, high cholesterol, or diabetes, and explore associations between bowel and bladder function and nutrition. This study will require 3 in person visits that are about 3 months apart. The total length of the study is about 6 months and includes 3 months of telenutrition counseling.

DETAILED DESCRIPTION:
The first phase of this study will include screening the participants' medical record for study eligibility. If potentially eligible, participants will partake in a secondary in-person screening assessment involving a fasting blood draw and weight, height, body fat, and waist circumference measurements. After the team receives the screening results and if participants continue to remain eligible, the second phase of the study (described below) will begin.

Following screening, participants will be enrolled into the 6-month study. Half of the enrolled participants will be scheduled for telenutrition counselling within the first three months of the study period. This group is called the "immediate treatment group". The other half will receive telenutrition counselling in the second three-month period. This group is called the "delayed treatment group". Participants will be informed which group they are assigned to and provided with details of the care that they will receive shortly after the screening phase is completed. Participants will have 50% chance of being assigned to the immediate treatment group and 50% chance of being assigned to the delayed treatment group.

Both groups will receive the same nutrition education and individualized nutrition counselling via videoconferencing with iPad FaceTime, which is aimed to decrease the risk of complications like obesity, high cholesterol, or diabetes, and explore associations between bowel and bladder function and nutrition. The telenutrition counselling consists of 6 sessions that are scheduled approximately 2 weeks apart. The first session will last approximately 1 hour, while sessions 2-6 will last approximately 30mins. During these sessions, the Registered Dietitian will share nutrition education tailored towards people with SCI. Participants will be involved in developing personal nutrition goals and the dietitian will help address barriers to meeting goals and provide individualized feedback to improve and maintain their nutrition. Telenutrition appointments will maintain privacy and will not be recorded.

To help participate in telenutrition sessions and complete the required assessments, each participant will receive an iPad mini with a 6-month data plan. Once study participation is complete, the investigators will stop the data plan but participants will get to keep the iPads. There are 3 outcome assessment spaced 3 months apart (baseline, short-term, and intermediate term). Each will include the same outcome assessments involving surveys, body measurements, and a blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with traumatic SCI
2. At least 1-year post-injury
3. Age 20 years of age or older
4. BMI > 22 kg/m2 at enrollment
5. Proficiency in English or Spanish
6. Living at home or in a private home setting (i.e., not an extended care facility) in the state of California
7. Able / willing to come to SCVMC for in-person assessments
8. Primarily a wheelchair user (>40 hours per week)
9. Able to use, or learn how to use, an iPad
10. Possess adequate decision-making capacity to provide independent informed consent

Exclusion Criteria:

1. Medical instability (e.g., uncontrolled hypertension, pneumonia, severe pressure injury)
2. Current self-reported pregnancy
3. Other medical condition requiring a strict specialized diet (e.g., renal failure, diabetes)
4. Participation in another diet program (e.g., Jenny Craig, Weight Watchers, clinic-based program) and/or participated in another diet program within the past 6 months
5. Current or past diagnosis of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating disorder)
6. Receiving enteral nutrition
7. Individuals without a primary care physician
8. HbA1c >7% (these individuals would need to be treated with metformin or other anti-diabetic medication and the intervention would have to be significantly altered for them)
9. Individuals who are in law enforcement custody

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Healthy Eating Index (HEI) scores | 0, 3 and 6 months
  HEI scores from participants' individual dietary intakes at different time-points of evaluations (baseline/pre-intervention, end of 3 months from baseline, end of 6 months from baseline) will be reported. Changes in HEI scores following intervention will be compared to pre-intervention baseline scores (within group comparison) as well as scores from the waitlisted group (between group comparison) and reported accordingly. In addition, longer-term changes in HEI scores (for individuals from the immediate intervention group) during the durability phase will also be reported.

SECONDARY OUTCOMES:
Blood lipid profile | 0, 3 and 6 months
  Lipid profile constituting of Triglycerides (TG), Total Cholesterol (TC); low-density lipoprotein (LDL) and High-density lipoprotein (HDL)- values (all expressed as mg/dL) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). In addition, absolute changes in values will also be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
HbA1C | 0, 3 and 6 months
  Blood values of HbA1C (expressed as percentage) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). Changes in percent values will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
Vitamin D | 0, 3 and 6 months
  Blood values of Vitamin D (expressed as ng/mL) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). In addition, absolute changes will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
high-sensitivity C-reactive protein [hs-CRP] | 0, 3 and 6 months
  Blood values of hs-CRP (expressed as mg/L) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). In addition, absolute changes will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group)
Body Mass Index (BMI) | 0, 3 and 6 months
  Multiple measures (weight in kg and height in meters) will be aggregated to arrive at one reported BMI values (expressed as kg/m^2). BMI values will be reported at all time-points of evaluations (baseline, end of 3 months and at the end of 6 months). Absolute changes in values will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
Waist circumference | 0, 3 and 6 months
  Waist circumference (in inches) will be reported at all time-points of evaluations (baseline, end of 3 months and at the end of 6 months). Absolute changes in values will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
Fat percent | 0, 3 and 6 months
  Fat percent (%) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). Changes in percentage values will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
Bowel function | 0, 3 and 6 months
  Changes in bowel function (as determined by the Simon Fraser University (SFU) bowel survey questions based on a rating scale) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). Changes in perceived rating will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
Bladder function | 0, 3 and 6 months
  Changes in bladder function (as determined by the SF-Qualiveen survey expressed as a score) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). Changes in scores will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
Quality of Life (Qol) measure | 0, 3 and 6 months
  Changes in Qol [using the Satisfaction With Life Scale (SWLS) survey based on a rating scale) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). Changes in perceived ratings will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).
Frequency of Autonomic Dysreflexia (AD) | 0, 3 and 6 months
  Changes in frequency of AD (as determined by the SFU AD survey questions expressed on a 5-point likert scale) will be reported at all time-points of evaluations (baseline/pre-intervention, end of 3 months and at the end of 6 months). Changes in rating will be reported following intervention compared to pre-intervention levels (within group comparison) and waitlisted group (between group comparison) as well as during the durability phase (for the immediate intervention group).

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Shem, MD, Principal Investigator — Santa Clara Valley Medical Center
Locations (1):
- Santa Clara Valley Medical Center, San Jose, California, United States